CLINICAL TRIAL: NCT03825601
Title: PET with [18F]Flumazenil As an Index of Neurodegeneration in MS: Sensitivity At an Early Disease Stage and Pathophysiological Meaning
Brief Title: PET with [18F]Flumazenil As an Index of Neurodegeneration in MS
Acronym: FLUMA-SEP-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C16-31
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis
Keywords: Patients,; Multiple Sclerosis,; Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with multiple sclerosis (Other): The multiple sclerosis group (n=30) will be subdivided in two subgroups: 15 patients with a relapsing remmitting MS (RRMS), and 15 patients with a primary progressive MS (PPMS).
  Interventions: Diagnostic Test: PET with [11C]Flumazenil
- healthy subjects (Other): 15 healthy subjects will be included. Among them 7 to 8 subjects will be matched for age and gender with the RRMS subgroup, and 7 to 8 will be matched for age and gender with the PPMS subgroup.
  Interventions: Diagnostic Test: PET with [11C]Flumazenil

INTERVENTIONS:
Diagnostic Test: PET with [11C]Flumazenil — 7T MRI sequences : TSE, T2w FLAIR GRE-T2* and DIR 3T MRI sequences: T1, T2, T1 with gadolinium, magnetization transfer, diffusion weighted, resting state fMRI.
  Other Names: 7T and 3T MRI

SUMMARY:
Beyond white matter pathology, grey matter damage is considered as a key player in disability onset and progression in Multiple Sclerosis (MS). The underlying substratum of grey matter damage is complex and pluriform, ranging from cortical demyelinating lesions, synapse and dendrite disappearance to neuronal cell death. Current Magnetic Resonance Imaging MRI techniques fail to fully assess and quantify grey matter pathology in this disease. The development of a quantitative marker of neurodegeneration for MS patients would allow: (i) to better understand the pathophysiological mechanisms underlying the distinct forms of MS; (ii) to stratify patients according to their prognosis; and (iii) to evaluate new therapies aimed at promoting neuroprotection. would allow to better understand the mechanisms underlying the distinct forms of MS, to stratify patients according to their prognosis, and to evaluate new therapies aimed at promoting neuroprotection.

DETAILED DESCRIPTION:
The investigators have recently shown that PET (Tomographie par Émission de Positrons) with [11C]Flumazenil ([11C]FMZ), that binds to the benzodiazepine site of GABA-A receptors, allowed to quantify and map neuronal damage in MS patients.

In the present project, the investigators will assess neuronal damage in MS using PET with [18F]Flumazenil ([18F]FMZ), at the early phase of either relapsing or primary progressive MS, and investigate the pathophysiological meaning of this neuronal damage by combining PET with Flumazenil with MRI at 7T and 3T.

The main objective will be to quantify and map [18F]FMZ binding changes in the grey matter of MS patients compared to controls, both at the group and the individual level. Secondary and exploratory objectives will be to investigate the relationship between Flumazenil binding changes and: i) cortical demyelinating lesions identified by several 7T MRI sequences ; ii) dendritic arborisation assessed by 3T DWI; ii) available MRI metrics obtained on a clinical 3T scan (grey matter atrophy MTR modifications, resting state connectivity); iv) clinical metrics.

This study will develop and assess a new imaging biomarker that has the potential to be used as an index of neurodegeneration in MS.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:

  * Aged 18-55 years old
  * Diagnosis of RRMS or PPMS according to the 2010 Mc Donald criteria
  * Disease duration < 10 years
  * Able to understand the study objective and procedure
  * Efficient contraception for women of potential child-bearing
  * Inscription to the national health care system
  * Having signed the written consent form
  * No current benzodiazepine or other GABAA-interacting drug (that have to be stopped 15 days before inclusion)
  * Accept to be informed of any incidental finding on imaging acquisitions
* Healthy subjects

  * Aged 18-55 years old
  * No evolutive pathology
  * Able to understand the study objective and procedure
  * Efficient contraception for women of potential child-bearing
  * Inscription to the national health care system
  * Having signed the written consent form
  * No concurrent benzodiazepine or other GABAA-interacting drug treatment (that have to be stopped 15 days before inclusion)
  * Accept to be informed of any incidental finding on imaging acquisitions

Exclusion Criteria:

* Any reason, which does not allow to perform MRI, including claustrophobia, the implant of a pace-maker or the presence of an intra-ocular foreign body.
* For women: pregnancy, lactation, lack of efficient contraception. A positive pregnancy test conducted at visit 2 will lead to the immediate exclusion of the subject.
* Current symptoms of severe or uncontrolled renal, hepatic, hematological, gastrointestinal pulmonary or cardiac disease.
* Radiation exposure during the last year before inclusion due to prior participations to other research protocols
* Other chronic neurological diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Concentration of benzodiazepine receptors (BZR) measured from 11C -Flumazenil binding in different groups | [0-2] MONTHS
  11C -Flumazenil binding in the grey matter : Concentration of benzodiazepine receptors (BZR) measured from 11C -Flumazenil binding kinetic analysis, and expressed as a Bmax estimation, in the cortex and deep grey matter of subjects.

SECONDARY OUTCOMES:
individual maps of neurodegeneration: changes in individual mapping of Flumazenil binding in different groups | [0-2] MONTHS
  Individual mapping of Flumazenil binding changes in the grey matter of patients with MS compared to healthy controls at the voxel level
volume of cortical lesions assessed on 7T MRI in different groups assessed in Cortical lesion volume | [0-2] MONTHS
  volume of cortical lesions assessed on 7T MRI in different groups assessed in Cortical lesion volume
volume of white matter lesions segmented on 3T T2 sequences: white matter lesion load | [0-2] MONTHS
  volume of white matter lesions segmented on 3T T2 sequences: white matter lesion load
Volume of gadolinium-enhanced white matter lesions on T1 sequence | [0-2] MONTHS
  Volume of gadolinium-enhanced white matter lesions assessed on T1 sequence
Voxel wise assessment of Magnetization transfer ratio (MTR) to assess changes in the grey and in the white matter in different groups | [0-2] MONTHS
  Voxel wise assessment of Magnetization transfer ratio (MTR) to assess changes in the grey and in the white matter in different groups
functional connectivity changes in patients | [0-2] MONTHS
  functional connectivity assessed on resting state fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique de Neuroscience, Groupe Hospitalier Pitié Salpêtrière, ICM, Pitié Salpêtrière, Paris, France